CLINICAL TRIAL: NCT04944589
Title: Comparison of Post-operative Pain Frequency in Non-vital Teeth After Single Visit Root Canal Versus Multiple Visit Root Canal Treatment
Brief Title: Comparison of Post-operative Pain Frequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hma Tanvir, Principal Investigator, Fatima Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14345
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Pain, Postoperative
Keywords: Endodontics, Non-vital teeth, Post-operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: : This study was a randomized controlled trial conducted at Department of Operative Dentistry, Fatima Memorial Hospital, Lahore, over a period of six months. A total of 302 patients presented with pulp necrosis in mandibular and maxillary first and second molar were included in this study and divided in two groups of 151. RCT of Group A patients was performed in single visit and RCT of group B patients was performed in multiple visits
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single visit root canal treatment(RCT) (Experimental): RCT(ROOT CANAL TREATMENT) of this group was performed in single visit including access cavity, chemo-mechanical preparation and obturation, all were done in one visit
  Interventions: Procedure: ROOT CANAL TREATMENT
- Multiple visit root canal treatment(RCT) (Experimental): RCT(ROOT CANAL TREATMENT) of this group was performed in multiple visit including access cavity, chemo-mechanical preparation and obturation, all were done in two or three visits
  Interventions: Procedure: ROOT CANAL TREATMENT

INTERVENTIONS:
Procedure: ROOT CANAL TREATMENT — Clinical endodontics involved in the goal of preventing and treating microbial contamination of pulps comprises of a number of treatments. Root canal endodontic therapy has one specific set of aims: to cure or prevent peri-radicular periodontitis, to conserve their natural teeth in function and aesthetics.

SUMMARY:
The objective of this study is:

* To compare the post-operative pain frequency after single visit root canal versus multiple visit root canal treatment in patients with non-vital teeth
* Post-operative pain is less frequent after single visit root canal than multiple visit root canal treatment in patients with non-vital teeth.

DETAILED DESCRIPTION:
METHODOLOGY This Randomized control trial was done in Outdoor patients Department of Operative Dentistry at Fatima Memorial Hospital. Informed written consent was taken from all patients who were willing to participate in the study. Patients who were diagnosed with non-vital teeth were considered for this study. Socio-demographic data and symptoms were recorded, subjects were examined and relevant investigations (vitality tests and radiographs) carried out. The patients were randomly divided into two groups through lottery method. Group A the treatment was done in one visit while in group B treatment was completed in two visits.

The standard procedure for both groups at first visit was administration of local anesthesia (1.8ml 2% Lignocaine with 1:10000 epinephrine), standard access cavity preparation followed by rubber dam isolation and pulp extirpation. After the confirmation of canal patency and working length radiograph, canals were prepared with the combination of hand files and engine-driven rotary nickel-titanium files (DENTSPLY Maillefer, Ballaigues, Switzerland) following manufacturer's instructions. 17%Ethylenediaminetetraacetic acid (EDTA )gel was used as a lubricant. Irrigation was performed with 2.5% NaOCl after each instrument in all cases. At the first visit, all teeth were prepared to working length and dried with paper points. Canals in Group A were filled with protaper universal gutta-percha (DENTSPLY Maillefer) and calcium hydroxide based sealer and restored with permanent restorative material in the same visit. In Group B after the canal preparation non-setting calcium hydroxide paste was placed with a sterile dry cotton pellet in the canal and tooth was restored with a minimum of 3.0mm Cavit. Patients in Group 2 were recalled after 1 week and the obturation technique same as Group 1 was followed in the second visit. After obturation, the patients in both the groups were recalled after 48 hours and assessed using visual analogue scale regarding presence and absence of post-operative pain. A value of 0-1 on Visual Analogue Scale (VAS) scale was considered as absence of pain.

The data was entered and analyzed in the SPSS-20. For descriptive analysis, mean and standard deviation was reported for age. Percentage for male and female participants was presented for gender distribution. The incidence of post-operative pain for single visit root canal and multiple visit root canal was determined. A chi-square test was used to determine the frequency of post-operative pain in both groups. A P value of 0.05 or less was taken as significant. Data was stratified more scientific manner in Pakistani population. So, the results of this study would add to the literature about the better, time saving and less painful (ROOT CANAL TREATMENT)RCT strategy in term of post- operative pain management.

ELIGIBILITY:
Inclusion Criteria:

* • Patients within age range 20-40 years.

  * Male/Female
  * Mature permanent first and second molar teeth (maxillary and mandibular)
  * Non-vital teeth (As defined in operational definitions)

Exclusion Criteria:

* • Any contraindication to local anesthesia, e.g. known allergy

  * Pregnancy.
  * endodontic re-treatment cases
  * Any physical or mental condition that would prevent jaw opening for the time required to complete the treatment.
  * Local acute infection/periapical radiolucency (diagnosed clinically, radio graphically )

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients within age range 20-40 years
Enrollment: 302 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Comprision of Post-Operative pain Frequency | 6 months
  After obturation, the patients in both the groups were recalled after 48 hours and assessed using visual analogue scale regarding presence and absence of post-operative pain. A value of 0-1 on VAS scale was considered as absence of pain

CONTACTS AND LOCATIONS:
Overall Officials: Huma Tanvir, BDS, Principal Investigator — Fatima Memorial Hospital
Locations (1):
- Huma Tanvir, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No